CLINICAL TRIAL: NCT04176809
Title: Impact of Routine Assessment of Health-Related Quality of Life Coupled With Therapeutic Information on Compliance With Endocrine Therapy in Patients With Non-metastatic Breast Cancer
Brief Title: Health-Related Quality of Life Coupled With Therapeutic Information on Compliance to Endocrine Therapy in Breast Cancer
Acronym: COMPLIANCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-A01323-54
Record Dates: First submitted 2019-11-20; First posted 2019-11-25 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
Keywords: Health Related Quality of Life; Compliance; Endocrine Therapy; Therapeutic Information
MeSH Terms: conditions — Breast Neoplasms; Patient Compliance

STUDY DESIGN:
Intervention Model Description: Eligible patients who agree to participate will be randomized into two parallel arms (ratio 1:1) by the minimization technique with stratification by age, stage, presence or absence of comorbidities and type of endocrine therapy prescribed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental): The intervention will consist in an electronic measurement of HRQoL before each consultation with delivery scores to clinicians, who can discuss it with patients and coupled with therapeutic information. Patients will complete the EORTC-Quality of Life Questionnaire (QLQ)-C30 and the EORTC-QLQ-Breast (BR) 23 questionnaires using the CHES software before their consultation, via a touch pad or from their home via a secure web portal. Therapeutic information will consist on workshops on various themes. Only attendance Workshop 1 will be required, other workshops will be optional. The aim of workshop 1 is to inform patients about their ET and treatment benefits. Two additional optional workshops on nutrition (Workshop 2) and fatigue (Workshop 3) will be offered. This workshops will be collective. Every month, a letter encouraging patients to regularly take their medication will be sent. This letter will also include some tips on how to deal with some particular side effects of ET.
  Interventions: Other: Routine Assessment of HRQoL coupled with Therapeutic Information
- Control arm (No Intervention): Participants in the control arm will receive standard care. They will not undergo digital HRQoL collection, and therapeutic information workshops will not be proposed.

INTERVENTIONS:
Other: Routine Assessment of HRQoL coupled with Therapeutic Information — Participants will complete the EORTC-QLQ-C30 and EORTC-QLQ-BR23 questionnaires before their consultation via the CHES software. The scores will then be generated and provided to clinicians in a graphic form, describing scores course. Access to CHES web portal will also be open to participants outside consultation time points, to enable them to monitor HRQoL if necessary. Workshop 1, will help patients to recognize and react to the occurrence of possible adverse effects, and anticipate their occurrence through appropriate preventive means. In workshop 2, participants will have the opportunity to express their representations and experiences related to their diet and the consequences of disease and treatments on diet. In workshop 3, participants can describe their experiences of fatigue and how their life is affected by it. Moreover, they can identify possible causes and finally discuss solutions to better this symptom. Every month, a reminder letter will also be sent to participants.
  Arms: Interventional arm

SUMMARY:
Only 59% of women with breast cancer (BC) treated with Endocrine Therapy (ET) remain compliant one year upon initial prescription, despite its proven effectiveness in reducing recurrence and improving survival. Health-related quality of life (HRQoL) in BC has been widely studied and the positive effects of its routine evaluation on the improvement of communication between patients and medical staff and survival have been highlighted. Recently, a link between HRQoL and compliance with ET has been suggested, which would suggest a potential role for HRQoL assessment in improving compliance with ET. With the advent of digital technologies, electronic collection of HRQoL on a tablet is now possible. Since compliance is a multidimensional phenomenon, a multifaceted intervention is necessary to improve it. Thus, the investigators hypothesize that systematic HRQoL assessment (using a tablet, prior to each consultation, with delivery of scores to clinicians) coupled with therapeutic information could have an impact on 12-month compliance with ET in patients with non-metastatic BC.

DETAILED DESCRIPTION:
In this study, 342 women with non-metastatic hormone receptor positive breast cancer with an indication for treatment with endocrine therapy will be include. Participants will be recruited at Dijon cancer center (Georges Francois Leclerc- center) in France. This center is specialized in cancer management, therefore clinicians are experienced in patient's HRQoL evaluation and are accustomed to take this criterion into consideration in the routine patient management. The study will be proposed to eligible participants by their doctors (oncologists, surgeons, radiation oncologists). Participants will be included at the time of the first prescription of ET (at the end of the treatments by surgery +/- chemotherapy +/- radiotherapy). Once included, participants will be randomized (ratio 1:1) by minimization and stratified by: age, stage, type of ET prescribed and presence or not of comorbidities, in 2 arms. Participants will then be referred to the clinical research associates, whose role will be to collect participant data (clinical and sociodemographic) in both study arms and to instruct participants in the interventional arm on how to use the Computer-based Health Evaluation System (CHES) software. For participants who wish to access the platform from home, a login and password will also be provided. If needed, clinical research associates will also assist participants to complete HRQoL questionnaires. This information will be collected in the case report form, to take into account the social desirability bias. The intervention will consist of numerical HRQoL assessment using the CHES software before each consultation (with delivery of scores to clinicians) coupled with therapeutic information. HRQoL assessment will be performed at each visit. As the aim of this project is to integrate this intervention in daily clinical practice, it will be performed in agreement with patients' routine follow-up. Participants will complete the questionnaires prior to each consultation, either at home via access to the web portal within 24 hours before consultation, or at the time of consultation. During consultation physician will have access to the results immediately, via the secure web portal, and will be able to discuss them with the participant. Therapeutic information will consist on 3 workshops. Workshop 1, entitled "Understanding the Prescription" will provide information on ET and its benefits. Two additional optional workshops on nutrition and fatigue will also be offered. Every month, a letter encouraging participants to regularly take their medication will be sent. Participants in the control group will follow standard care. Both in two arms, HRQoL will be evaluated at baseline using the FACT-G questionnaire to ensure the comparability of groups concerning HRQoL at inclusion, and again at 12 months. HRQoL assessment will be performed using a traditional paper questionnaire and scores will not be provided to clinicians. Anxiety and depression, social support and participant satisfaction with care will also be assessed in both arms at baseline and 12 months after. Sociodemographic characteristics, medical and surgical history, date of tumor diagnosis, tumor characteristics, previous treatments, participant clinical characteristics at inclusion and at each follow-up visit (weight, height, overall patient condition), concomitant treatment, type of ET received, HRQoL data (FACT-G), anxiety and depression (HADS), social support (SSQ6), treatment modification (change in the type of ET), treatment-related toxicities and their grade will be collected. Participant satisfaction with provided care will be measured. Clinicians' perceptions of systematic HRQoL assessment will be collected via an ad hoc questionnaire. Sociodemographic data and reasons for refusing to participate will also be documented for patients who refuse to participate. Data on patients' withdrawal or death will be documented in the case report form. Reasons for study withdrawal should also be documented. All data from this study will be transcribed in an electronic case report form. A descriptive analysis of participants' clinical and socio-demographic characteristics at inclusion will be performed for each arm. All HRQoL scores will be calculated according to FACT-G guidelines and described according to the arm (interventional arm or control arm). A logistic regression model will be used to assess the capacity of HRQoL to predict 12-month compliance with endocrine therapy. The modulatory potential of social support on compliance will be assessed using an interaction term between the availability / satisfaction of social support that patients receive and HRQoL in a logistic regression model. The modulatory potential of psychological distress on compliance will be assessed using an interaction term between patient anxiety / depression and HRQoL in a logistic regression model.

An analysis of missing HRQoL data profiles will also be performed. If a Missing Not At Random (MNAR) profile is demonstrated / suspected, multiple imputation of missing data can be performed in sensitivity analysis, taking into account the variables associated with the occurrence of missing data. As a sensitivity analysis, the investigators will performed a contamination-based intent-to-treat analysis to account for potential cross-contamination between the arms.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 and over
* With non-metastatic hormone receptor positive breast cancer
* Women will have to be at the end of primary treatment
* An indication for endocrine therapy treatment during 5 to 10 years
* be affiliated to a French social security scheme or beneficiary of such a scheme
* agreed to participate by signing a written consent

Exclusion Criteria:

* Participants who participate in another clinical trial where HRQoL is assessed
* Women for whom HRQoL evaluation is not possible (cognitive disorders, psychiatric disorders, people who do not speak French, etc.).
* Vulnerable participants (pregnant women, etc.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2021-05-14 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants compliant with endocrine therapy as assessed by Morisky Green Levine (MGL) scale | 12 months after the onset of endocrine therapy
  Compliance with endocrine therapy, will be evaluated using the Morisky Green Levine scale (MGL). It has a range of 0 to 4, where 0 is very low and 4 is highest. Patients are categorized according to three levels of adherence: high (score equal to 4), moderate (score equal to 2 or 3) and low (score equal to 0 or 1). Participants will be considered as compliant if they have a high adherence score in MGL scale.

SECONDARY OUTCOMES:
Number of anxious and depress participants as assessed by Hospital Anxiety and Depression Scale (HADS) | at baseline and 12 months after the onset of endocrine therapy
  HADS has 14 items rated from 0 to 3 and covers 2 dimensions. Seven questions related to the anxiety dimension and seven other related to the depressive dimension, yielding 2 scores, A (Anxiety) and D (Depression). The maximum score for each dimension is 21. A score of 11 or higher indicates the probable presence of the disorder.
social support as assessed by Sarason's Social Support Questionnaire 6-item (SSQ6) | at baseline and 12 months after the onset of endocrine therapy
  Social support is measured across 2 dimensions: support availability, through the number of contacts that the patient can count on (0 to 9 people) and quality of support, through patient satisfaction with support received.
  Each item represents a situation in which the patient may need support. Patient is asked to cite the number of people that she could count on in that particular situation. Concerning the second item, the patient is asked to assess satisfaction with the support provided. The scores are generated according to Sarason's recommendations. A score is calculated for each dimension. Support availability score is calculated as the sum of the number of people available for the 6 items, this score ranges from 0 to 54, with 54 representing the highest availability. The social support satisfaction score is calculated by the sum of the satisfaction of the 6 items. This score ranges from 6 to 36, with 36 representing the highest level of satisfaction
HRQoL data using Functional Assessment Cancer Therapy-General questionnaire (FACT-G) | at baseline and 12 months after the onset of endocrine therapy
  HRQoL data using the Functional Assessment Cancer Therapy General (FACT-G) questionnaire will be assessed at inclusion in both arms to ensure comparability between groups and at 12 months, to assess the predictive value of HRQoL on compliance to endocrine therapy. The FACT-G instrument assesses 4 HRQoL domains: physical well-being (7 items); social and/or family well-being (7 items); emotional well-being (6 items); and functional well-being (7 items). Respondents use a 5-point Likert-type scale which rates the relevant domain from 0 (not at all) to 4 (very much). From these subscales a global score is obtained. The FACT-G total score vary from 0 to 108. The higher the score, the better the HRQoL.
Patient satisfaction with care as assessed by European Organization Research and Treatment Cancer 33-item Satisfaction with cancer care core questionnaire (EORTC PATSAT-C33) and its module 7-item Outpatient Satisfaction with care (EORTC OUT-PATSAT-7) | at baseline and 12 months after the onset of endocrine therapy
  The European Organization Research and Treatment Cancer 33-item Satisfaction with cancer care core (EORTC PATSAT-C33) questionnaire and its module 7-item Outpatient Satisfaction with care (EORTC OUT-PATSAT-7) assess perceptions of cancer patients regarding the quality of care received. The EORTC PATSAT-C33 includes 3 sections on the perceived quality of care provided by physicians, radiotherapy nurses/technicians and services/care organization. The first one includes 3 dimensions that address technical skills, quality and quantity of information exchanged and behavior. The second one has 2 dimensions: information provision and reactivity and affective behavior. The third one has 3 dimensions: coordination, interaction with the healthcare team and 5 single items. The module EORTC-OUT-PATSAT7 includes 2 dimensions dealing with convenience of care and transition and a single item on continuity of care. The score vary from 0 to 100. A higher score indicates higher level of satisfaction.
Physician perception regarding the utility of systematic HRQoL evaluation as assessed by an ad-hoc questionnaire | through study completion, an average of 3 years
  Physician perception regarding the utility of systematic HRQoL evaluation will be assessed using an ad hoc questionnaire derived from the work of Velikova, including the perceived utility and satisfaction of routine assessment HRQoL, reasons for use/non-use and the intention to adopt this assessment in routine care. This questionnaire does not generate a score but give us information on the points mention above.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle DESMOULINS, MD, Principal Investigator — Georges François Leclerc Centre
Locations (1):
- Centre Georges François Leclerc, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huiart L, Bardou VJ, Giorgi R. [The importance of adherence to oral therapies in the field of oncology: the example of breast cancer]. Bull Cancer. 2013 Oct;100(10):1007-15. doi: 10.1684/bdc.2013.1830. French. PMID 24113516
- [Background] Ayres LR, Baldoni Ade O, Borges AP, Pereira LR. Adherence and discontinuation of oral hormonal therapy in patients with hormone receptor positive breast cancer. Int J Clin Pharm. 2014 Feb;36(1):45-54. doi: 10.1007/s11096-013-9833-5. Epub 2013 Aug 11. PMID 23934310
- [Background] Hugtenburg JG, Timmers L, Elders PJ, Vervloet M, van Dijk L. Definitions, variants, and causes of nonadherence with medication: a challenge for tailored interventions. Patient Prefer Adherence. 2013 Jul 10;7:675-82. doi: 10.2147/PPA.S29549. Print 2013. PMID 23874088
- [Background] Egede LE, Gebregziabher M, Dismuke CE, Lynch CP, Axon RN, Zhao Y, Mauldin PD. Medication nonadherence in diabetes: longitudinal effects on costs and potential cost savings from improvement. Diabetes Care. 2012 Dec;35(12):2533-9. doi: 10.2337/dc12-0572. Epub 2012 Aug 21. PMID 22912429
- [Background] Cheung WY, Lai EC, Ruan JY, Chang JT, Setoguchi S. Comparative adherence to oral hormonal agents in older women with breast cancer. Breast Cancer Res Treat. 2015 Jul;152(2):419-27. doi: 10.1007/s10549-015-3455-7. Epub 2015 Jun 13. PMID 26070268
- [Background] Murphy CC, Bartholomew LK, Carpentier MY, Bluethmann SM, Vernon SW. Adherence to adjuvant hormonal therapy among breast cancer survivors in clinical practice: a systematic review. Breast Cancer Res Treat. 2012 Jul;134(2):459-78. doi: 10.1007/s10549-012-2114-5. Epub 2012 Jun 12. PMID 22689091
- [Background] Weaver KE, Camacho F, Hwang W, Anderson R, Kimmick G. Adherence to adjuvant hormonal therapy and its relationship to breast cancer recurrence and survival among low-income women. Am J Clin Oncol. 2013 Apr;36(2):181-7. doi: 10.1097/COC.0b013e3182436ec1. PMID 22314001
- [Background] Hsieh KP, Chen LC, Cheung KL, Chang CS, Yang YH. Interruption and non-adherence to long-term adjuvant hormone therapy is associated with adverse survival outcome of breast cancer women--an Asian population-based study. PLoS One. 2014 Feb 21;9(2):e87027. doi: 10.1371/journal.pone.0087027. eCollection 2014. PMID 24586261
- [Background] Taketani K, Tokunaga E, Yamashita N, Tanaka K, Akiyoshi S, Okada S, Ando K, Kimura Y, Saeki H, Oki E, Morita M, Kusumoto T, Maehara Y. Early discontinuation of adjuvant hormone therapy is associated with a poor prognosis in Japanese breast cancer patients. Surg Today. 2014 Oct;44(10):1841-6. doi: 10.1007/s00595-013-0762-7. Epub 2013 Oct 19. PMID 24142101
- [Background] Hadji P, Blettner M, Harbeck N, Jackisch C, Luck HJ, Windemuth-Kieselbach C, Zaun S, Kreienberg R. The Patient's Anastrozole Compliance to Therapy (PACT) Program: a randomized, in-practice study on the impact of a standardized information program on persistence and compliance to adjuvant endocrine therapy in postmenopausal women with early breast cancer. Ann Oncol. 2013 Jun;24(6):1505-12. doi: 10.1093/annonc/mds653. Epub 2013 Feb 1. PMID 23378537
- [Background] Ziller V, Kyvernitakis I, Knoll D, Storch A, Hars O, Hadji P. Influence of a patient information program on adherence and persistence with an aromatase inhibitor in breast cancer treatment--the COMPAS study. BMC Cancer. 2013 Sep 4;13:407. doi: 10.1186/1471-2407-13-407. PMID 24006873
- [Background] Markopoulos C, Neven P, Tanner M, Marty M, Kreienberg R, Atkins L, Franquet A, Gnant M, Neciosup S, Tesarova P, Barni S, Deschamp V. Does patient education work in breast cancer? Final results from the global CARIATIDE study. Future Oncol. 2015;11(2):205-17. doi: 10.2217/fon.14.179. PMID 25591836
- [Background] Hadji P. Improving compliance and persistence to adjuvant tamoxifen and aromatase inhibitor therapy. Crit Rev Oncol Hematol. 2010 Feb;73(2):156-66. doi: 10.1016/j.critrevonc.2009.02.001. Epub 2009 Mar 18. PMID 19299162
- [Background] Madan A, Borckardt JJ, Connell A, Book SB, Campbell S, Gwynette MF, Wimberly LA, Wagner M, Weinstein B, McLeod-Bryant S, Cooney H, Herbert J. Routine assessment of patient-reported outcomes in behavioral health: room for improvement. Qual Manag Health Care. 2010 Jan-Mar;19(1):70-81. doi: 10.1097/QMH.0b013e3181ccbc53. PMID 20042935
- [Background] Epplein M, Zheng Y, Zheng W, Chen Z, Gu K, Penson D, Lu W, Shu XO. Quality of life after breast cancer diagnosis and survival. J Clin Oncol. 2011 Feb 1;29(4):406-12. doi: 10.1200/JCO.2010.30.6951. Epub 2010 Dec 20. PMID 21172892
- [Background] Takada K, Kashiwagi S, Fukui Y, Goto W, Asano Y, Morisaki T, Takashima T, Hirakawa K, Ohira M. Prognostic value of quality-of-life scores in patients with breast cancer undergoing preoperative chemotherapy. BJS Open. 2018 Nov 26;3(1):38-47. doi: 10.1002/bjs5.50108. eCollection 2019 Feb. PMID 30734014
- [Background] Chu WO, Dialla PO, Roignot P, Bone-Lepinoy MC, Poillot ML, Coutant C, Arveux P, Dabakuyo-Yonli TS. Determinants of quality of life among long-term breast cancer survivors. Qual Life Res. 2016 Aug;25(8):1981-90. doi: 10.1007/s11136-016-1248-z. Epub 2016 Feb 25. PMID 26914102
- [Background] Lavdaniti M, Owens DA, Liamopoulou P, Marmara K, Zioga E, Mantzanas MS, Evangelidou E, Vlachou E. Factors Influencing Quality of Life in Breast Cancer Patients Six Months after the Completion of Chemotherapy. Diseases. 2019 Feb 24;7(1):26. doi: 10.3390/diseases7010026. PMID 30813488
- [Background] Velikova G, Booth L, Smith AB, Brown PM, Lynch P, Brown JM, Selby PJ. Measuring quality of life in routine oncology practice improves communication and patient well-being: a randomized controlled trial. J Clin Oncol. 2004 Feb 15;22(4):714-24. doi: 10.1200/JCO.2004.06.078. PMID 14966096
- [Background] Basch E, Deal AM, Kris MG, Scher HI, Hudis CA, Sabbatini P, Rogak L, Bennett AV, Dueck AC, Atkinson TM, Chou JF, Dulko D, Sit L, Barz A, Novotny P, Fruscione M, Sloan JA, Schrag D. Symptom Monitoring With Patient-Reported Outcomes During Routine Cancer Treatment: A Randomized Controlled Trial. J Clin Oncol. 2016 Feb 20;34(6):557-65. doi: 10.1200/JCO.2015.63.0830. Epub 2015 Dec 7. PMID 26644527
- [Background] Denis F, Lethrosne C, Pourel N, Molinier O, Pointreau Y, Domont J, Bourgeois H, Senellart H, Tremolieres P, Lizee T, Bennouna J, Urban T, El Khouri C, Charron A, Septans AL, Balavoine M, Landry S, Solal-Celigny P, Letellier C. Randomized Trial Comparing a Web-Mediated Follow-up With Routine Surveillance in Lung Cancer Patients. J Natl Cancer Inst. 2017 Sep 1;109(9). doi: 10.1093/jnci/djx029. PMID 28423407
- [Background] Pinheiro LC, Wheeler SB, Reeder-Hayes KE, Samuel CA, Olshan AF, Reeve BB. Investigating Associations Between Health-Related Quality of Life and Endocrine Therapy Underuse in Women With Early-Stage Breast Cancer. J Oncol Pract. 2017 May;13(5):e463-e473. doi: 10.1200/JOP.2016.018630. Epub 2017 Mar 14. PMID 28291383
- [Background] Kotronoulas G, Kearney N, Maguire R, Harrow A, Di Domenico D, Croy S, MacGillivray S. What is the value of the routine use of patient-reported outcome measures toward improvement of patient outcomes, processes of care, and health service outcomes in cancer care? A systematic review of controlled trials. J Clin Oncol. 2014 May 10;32(14):1480-501. doi: 10.1200/JCO.2013.53.5948. Epub 2014 Apr 7. PMID 24711559
- [Background] Ruland CM, Andersen T, Jeneson A, Moore S, Grimsbo GH, Borosund E, Ellison MC. Effects of an internet support system to assist cancer patients in reducing symptom distress: a randomized controlled trial. Cancer Nurs. 2013 Jan-Feb;36(1):6-17. doi: 10.1097/NCC.0b013e31824d90d4. PMID 22495503
- [Background] Eggersmann TK,Harbeck N, Schinkoethe T, Riese C. eHealth solutions for therapy management in oncology. Breast Cancer Manag. 2018; 6(3):101-106.
- [Background] Holzner B, Giesinger JM, Pinggera J, Zugal S, Schopf F, Oberguggenberger AS, Gamper EM, Zabernigg A, Weber B, Rumpold G. The Computer-based Health Evaluation Software (CHES): a software for electronic patient-reported outcome monitoring. BMC Med Inform Decis Mak. 2012 Nov 9;12:126. doi: 10.1186/1472-6947-12-126. PMID 23140270
- [Background] Osoba D, Rodrigues G, Myles J, Zee B, Pater J. Interpreting the significance of changes in health-related quality-of-life scores. J Clin Oncol. 1998 Jan;16(1):139-44. doi: 10.1200/JCO.1998.16.1.139. PMID 9440735
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Fayers PM, Aaronson NK, Bjordal K, Groenvold M, Curran D, Bottomley A, on behalf of the EORTC Quality of Life Group. The EORTC QLQ-C30 Scoring Manual (3rd Edition).2001.
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130
- [Background] Lepine JP, Godchau M, Brun P. Anxiety and depression in inpatients. Lancet. 1985 Dec 21-28;2(8469-70):1425-6. doi: 10.1016/s0140-6736(85)92589-9. No abstract available. PMID 2867417
- [Background] Costet N, Lapierre V, Benhamou E, Le Gales C. Reliability and validity of the Functional Assessment of Cancer Therapy General (FACT-G) in French cancer patients. Qual Life Res. 2005 Jun;14(5):1427-32. doi: 10.1007/s11136-004-5531-z. PMID 16047518
- [Background] Conroy T, Mercier M, Bonneterre J, Luporsi E, Lefebvre JL, Lapeyre M, Puyraveau M, Schraub S. French version of FACT-G: validation and comparison with other cancer-specific instruments. Eur J Cancer. 2004 Oct;40(15):2243-52. doi: 10.1016/j.ejca.2004.06.010. PMID 15454249
- [Background] Bredart A, Anota A, Young T, Tomaszewski KA, Arraras JI, Moura De Albuquerque Melo H, Schmidt H, Friend E, Bergenmar M, Costantini A, Vassiliou V, Hureaux J, Marchal F, Tomaszewska IM, Chie WC, Ramage J, Beaudeau A, Conroy T, Bleiker E, Kulis D, Bonnetain F, Aaronson NK; EORTC Quality of Life Group. Phase III study of the European Organisation for Research and Treatment of Cancer satisfaction with cancer care core questionnaire (EORTC PATSAT-C33) and specific complementary outpatient module (EORTC OUT-PATSAT7). Eur J Cancer Care (Engl). 2018 Jan;27(1). doi: 10.1111/ecc.12786. Epub 2017 Nov 2. PMID 29094784
- [Background] Rascle N, Bruchon-Schweitzer M, Sarason IG. Short form of Sarason's Social Support Questionnaire: French adaptation and validation. Psychol Rep. 2005 Aug;97(1):195-202. doi: 10.2466/pr0.97.1.195-202. PMID 16279325
- [Background] Bruchon-Schweitzer M. Psychologie de la santé. Modèles, concepts et méthodes. 1er éd. Paris : Dunod. 2002A.
- [Background] Velikova G, Keding A, Harley C, Cocks K, Booth L, Smith AB, Wright P, Selby PJ, Brown JM. Patients report improvements in continuity of care when quality of life assessments are used routinely in oncology practice: secondary outcomes of a randomised controlled trial. Eur J Cancer. 2010 Sep;46(13):2381-8. doi: 10.1016/j.ejca.2010.04.030. Epub 2010 Jun 1. PMID 20570138
- [Derived] Mamguem Kamga A, Di Martino C, Anota A, Paget-Bailly S, Coutant C, Arveux P, Desmoulins I, Dabakuyo-Yonli TS. Impact of routine assessment of health-related quality of life coupled with therapeutic information on compliance with endocrine therapy in patients with non-metastatic breast cancer: protocol for a randomized controlled trial. Trials. 2020 Jun 16;21(1):527. doi: 10.1186/s13063-020-04397-w. PMID 32546198